CLINICAL TRIAL: NCT00003563
Title: Phase III Randomized Trial of Gadolinium Texaphyrin (PCI-0120) Injection as a Radiation Sensitizer in Patients Receiving Whole Brain Radiation Therapy for the Treatment of Brain Metastases
Brief Title: Radiation Therapy Plus Gadolinium Texaphyrin in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066627; PCI-P120-9801; MSKCC-00088; UCLA-9808021; NCI-V98-1470
Record Dates: First submitted 1999-11-01; First posted 2004-04-30 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2008-06

CONDITIONS: Metastatic Cancer
Keywords: tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms

ARMS (2):
- WBRT (Experimental): 3 Gy of WBRT daily for a total of 10 days
  Interventions: Radiation: WBRT
- MGd (Experimental): IV does of 5.0 mg/kg MGd plus WBRT
  Interventions: Radiation: WBRT; Drug: MGd

INTERVENTIONS:
Radiation: WBRT — 3 GY of WBRT daily for a total of 10 days
Drug: MGd — 5.0 mg /kg MGd plus WBRT
  Other Names: MGd plus WBRT
  Arms: MGd

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Gadolinium texaphyrin may increase the effectiveness of radiation therapy by making tumor cells more sensitive to radiation. It is not yet known whether giving gadolinium texaphyrin with radiation therapy is more effective than radiation therapy alone in treating brain metastases.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without gadolinium texaphyrin in treating patients who have brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of gadolinium texaphyrin administered prior to whole brain radiotherapy in patients with brain metastases. II. Compare the efficacy and toxicity of whole brain radiotherapy with or without gadolinium texaphyrin in these patients. III. Assess the quality of life of these patients.

OUTLINE: This is a randomized, two stage, multicenter study. Patients are stratified according to RTOG recursive partitioning analysis class (RPA class 1 vs class 2) and tumor type (breast vs lung vs other). Stage 1 (lead-in): All patients receive gadolinium texaphyrin IV over 5-10 minutes on the 10 days that they receive radiotherapy. Approximately 2-5 hours later, patients undergo whole brain radiotherapy. Stage 2 (randomization): Patients are randomized to one of two treatment arms. Patients in arm I undergo whole brain radiotherapy for 10 days. Patients in arm II receive gadolinium texaphyrin and radiotherapy as in stage 1. Quality of life is assessed on days 10 and 28, then monthly for 5 months, and then every 3 months thereafter. Patients are followed at day 28, then monthly for 5 months, and then every 3 months until death.

PROJECTED ACCRUAL: The lead-in phase will accrue at least 25-30 patients and the randomization phase will accrue 400 patients (200/arm) over a 12 month period.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven solid tumor with parenchymal brain metastasis Solitary metastasis eligible only if refused surgery or surgical resection deemed inappropriate No leptomeningeal metastases or subarachnoid spread of tumor No small cell lung cancer, germ cell tumors, lymphoma, or leukemia No liver metastases, unless from breast cancer No more than 1 site of extracranial metastases (multiple bone or lung metastases count as one site), unless from breast cancer Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 50,000/mm3 Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) AST and ALT no greater than 2 times ULN Renal: Creatinine no greater than 2.0 mg/mL Other: No history of porphyria No history of G6PD deficiency HIV negative No other major medical illnesses No major psychiatric impairment Not pregnant or nursing Negative pregnancy test

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No chemotherapy during and for 2 weeks after gadolinium texaphyrin therapy Endocrine therapy: Concurrent hormonal therapy allowed Radiotherapy: No prior cranial radiation, including prior stereotactic radiosurgery No plan for radiosurgery or radiation boost following whole brain radiotherapy Concurrent radiotherapy allowed to other sites, except kidneys and liver Surgery: No prior subtotal or total resection of brain metastases (except biopsies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 1998-08; Primary Completion 2001-09 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Renschler, MD, Study Chair — Pharmacyclics LLC.
Locations (35):
- United States (31):
  - Marin Oncology Associates, Inc., Greenbrae, California
  - Kaiser Permanente Medical Group, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Charlotte County Radiation Therapy Regional Center, Port Charlotte, Florida
  - Emory Clinic, Atlanta, Georgia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Hematology and Oncology Services - Metairie, Metairie, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Harper Hospital and Wayne State University, Detroit, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - North Memorial Research Center, Minneapolis, Minnesota
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New Mexico Oncology-Hematology, Albuquerque, New Mexico
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abington Hematology Oncology Associates, Meadowbrook, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Presbyterian-University Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec

REFERENCES:
- [Result] Li J, Bentzen SM, Li J, Renschler M, Mehta MP. Relationship between neurocognitive function and quality of life after whole-brain radiotherapy in patients with brain metastasis. Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):64-70. doi: 10.1016/j.ijrobp.2007.09.059. PMID 18406884
- [Result] Li J, Bentzen SM, Renschler M, Mehta MP. Regression after whole-brain radiation therapy for brain metastases correlates with survival and improved neurocognitive function. J Clin Oncol. 2007 Apr 1;25(10):1260-6. doi: 10.1200/JCO.2006.09.2536. PMID 17401015